CLINICAL TRIAL: NCT05830110
Title: Patterned Multichannel Vibrotactile Stimulation for the Longitudinal Treatment of Moderate Stage Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synergic Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VCR-Longitudinal
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease
Keywords: vibrotactile
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will serve as their own control, receiving alternating active and sham therapy at two-month intervals.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active vibrotactile coordinated reset (Active Comparator): mechanical vibrotactile stimulation to the fingers in a defined pattern
  Interventions: Device: Active Vibrotactile Coordinated Reset
- Sham vibrotactile coordinated reset (Sham Comparator): mechanical vibrotactile stimulation to the fingers in a defined pattern
  Interventions: Device: Sham vibrotactile coordinated reset

INTERVENTIONS:
Device: Active Vibrotactile Coordinated Reset — Gloves providing vibrotactile coordinated reset stimulation
  Arms: Active vibrotactile coordinated reset
Device: Sham vibrotactile coordinated reset — Gloves providing sham vibrotactile coordinated reset stimulation
  Arms: Sham vibrotactile coordinated reset

SUMMARY:
The purpose of the present research is to examine the effectiveness of a non-invasive, vibrotactile stimulation protocol, known as coordinated reset (CR), for the alleviation of motor symptoms in patients with Parkinson's disease (PD). PD patients exhibit rigidity, slowness (bradykinesia) and poverty (akinesia) of movement as well as other symptoms. Treatment for PD is either pharmacological (first line) or invasive deep brain stimulation. The non-invasive, vibrotactile stimulation approach uses a novel stimulation pattern to disrupt the pathophysiological mechanism that is responsible for PD symptoms and thus restore motor function.

DETAILED DESCRIPTION:
Up to thirty adults with bilateral, moderate stage idiopathic PD will be enrolled in this longitudinal study. Participants will serve as their own control, receiving alternating active and sham therapy at two-month intervals. This longitudinal protocol will be open-ended to enable continued treatment to those interested / motivated.

Study treatment will consist of daily, four-hour vibrotactile Coordinated Reset (vCR) stimulation sessions on a continual basis. All daily vCR stimulation sessions will occur at the participant's home (ON-medication) and can be broken up into two, two-hour blocks (with no more than 12 hours between stimulation blocks) to be less cumbersome and better integrate into the participant's daily life. Daily home-based treatment will be unsupervised, though timely support is guaranteed by Synergic Medical Technologies (SMT) support staff when needed (e.g., when usability or IT issues arise). Daily stimulation / device usage will be automatically logged by the device and continuously monitored by SMT staff, meanwhile participants will keep a med diary so we can monitor their med usage (and how it relates to extended exposure) over time. Participants will be able to transition to an as-needed basis with treatment after four months and once they are familiar with the treatment and their body's response to it, to better alleviate PD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* between the ages 45 and 90
* diagnosis of bilateral, moderate stage idiopathic PD
* qualify for EEG procedures

Exclusion Criteria:

* on dopamine agonist medications and exhibiting compulsive behaviors

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society - Change in Universal Parkinson Disease Rating Scale (MDS-UPDRS) | baseline, 2 months, 4 months
  Change in MDS-UPDRS score using Part 3 of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Phan Luu, PhD, Principal Investigator — Synergic Medical Technologies, Inc.
Locations (1):
- Synergic Medical Technologies, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No